CLINICAL TRIAL: NCT01819909
Title: Prospective Randomized Trial of Rotator Cuff Repair Postoperative Rehabilitation: Jackins' Exercises Versus Pulleys
Brief Title: Effectiveness Study of Postoperative Rotator Cuff Repair Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Orthopedic Institute, Sioux Falls, SD (Other)
Responsible Party: Principal Investigator, Keith Baumgarten, MD, Orthopedic Institute, Sioux Falls, SD
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Jackins
Record Dates: First submitted 2012-12-23; First posted 2013-03-28 (Estimated); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Full Thickness Rotator Cuff Tear
Keywords: Rotator cuff repair; Shoulder; Surgery; Rehabilitation; Pulleys; Jackins

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Postoperative Jackins Exercise Protocol (Experimental): Jackin's exercises were initially designed for patients with difficulty performing forward elevation. The patient initially is positioned supine to perform shoulder flexion. When the patient can actively elevate in the supine position, one to two pounds of weight is placed in the patients hand and the patient is asked to repeat the maneuver of supine active elevation. When the patient can do this with little difficulty, the head of the bed is elevated approximately 20 degrees from the supine position and the sequence is repeated. Once the patient is able to perform flexion in this elevated head position, the inclination of the patient is increased in 20 degree increments until the patient is able to perform upright sitting shoulder flexion.
  Interventions: Procedure: Postoperative Jackins Exercise Protocol
- Postoperative Pulleys Exercise Protocol (Experimental): Pulleys have been used in postoperative shoulder rehabilitation to improve passive as well as active range of motion and develop strength.
  Interventions: Procedure: Postoperative Pulleys Exercise Protocol

INTERVENTIONS:
Procedure: Postoperative Jackins Exercise Protocol — Jackin's exercises were initially designed for patients with difficulty performing forward elevation. The patient initially is positioned supine to perform shoulder flexion. When the patient can actively elevate in the supine position, one to two pounds of weight is placed in the patients hand and the patient is asked to repeat the maneuver of supine active elevation. When the patient can do this with little difficulty, the head of the bed is elevated approximately 20 degrees from the supine position and the sequence is repeated. Once the patient is able to perform flexion in this elevated head position, the inclination of the patient is increased in 20 degree increments until the patient is able to perform upright sitting shoulder flexion.
  Arms: Postoperative Jackins Exercise Protocol
Procedure: Postoperative Pulleys Exercise Protocol — Pulleys have been used in postoperative shoulder rehabilitation to improve passive as well as active range of motion and develop strength.
  Arms: Postoperative Pulleys Exercise Protocol

SUMMARY:
There are very few level 1 or level 2 evidence studies that examine postoperative rehabilitation of rotator cuff repair and shoulder arthroplasty. A systematic review of level 1 or level 2 evidence studies was performed (Baumgarten et al., Sports Health, 2009) that found only four studies that examined rotator cuff repair rehabilitation.

The current study was performed to determine if there is a significant difference in passive glenohumeral joint range of motion, active glenohumeral joint range of motion, scapular substitution, and subjects measured outcome scores (clinimetrics) in patients who undergo rotator cuff repair when treated postoperatively with pulley exercises compared to Jackins' exercises.

Null Hypothesis: There will be no significant difference in passive range of motion, active range of motion, scapular substitution, and subject measured outcomes scores in subjects who undergo rotator cuff repair when treated with pulley exercises compared to Jackins' exercises.

DETAILED DESCRIPTION:
Scapulothoracic substitution for forward elevation is seen clinically when patients have shoulder pain. The patient uses the trapezius musculature to superiorly elevate the upper extremity instead of using the deltoid and the rotator cuff for upper extremity elevation. Scapulothoracic substitution does not occur in healthy shoulders. Excessive scapular movement can be due to an attempt to substitute for poorly functioning shoulder musculature or tightness of the capsular structures of the glenohumeral joint.

Pulleys have been used in postoperative shoulder rehabilitation to improve passive as well as active range of motion and develop strength. Jackins described a series of exercises that are used to improve active range of motion and develop strength without the use of pulleys. The use of pulleys in the post-operative care for patients who have had shoulder surgery is thought to contribute to excessive scapular motion. To date, there has not been any study that compares the use of pulleys and Jackins' exercises with respect to active range of motion, scapulothoracic substitution, and objective patient outcomes measures. Due to the lack of level 1 or 2 evidence postoperative rehabilitation studies, a prospective randomized study should be performed on patients that have underwent rotator cuff repair.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing post-operative rehabilitation for a rotator cuff repair

Exclusion Criteria:

* Patients who do not have permission from their treating surgeon to enroll in this study.

Patients who have undergone a previous rotator cuff repair on the non-operated side.

Patients who have undergone a previous rotator cuff repair on the ipsilateral shoulder.

Patients who have a history of adhesive capsulitis. Patients who are unwilling to participate in all aspects of the study. Patients who are cognitively impaired. Patients with known axillary or suprascapular neuropathy. Patients with a painful or dysfunctional contralateral shoulder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2008-11 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Change in Western Ontario Rotator Cuff Index (WORC) | Baseline, 6 weeks, 12 weeks, 6 months, 1 year
  The WORC(ref 6) is a valid,reliable, and responsive patient-reported outcomes measures that assesses response to treatment for rotator cuff disease. A minimally important clinical difference (MCID) has been determined. Its use has been recommended in clinical trials.

SECONDARY OUTCOMES:
Change in scapular substitution (centimeters) | Baseline, 6 weeks, 12 weeks, 6 months, 1 year
  A novel technique for measuring scapular substitution has been developed by the investigators of this study (Baumgarten et al. Int J Sports Phys Ther. 2012; 7: 39-48).
Change in range of motion (degrees) | Baseline, 6 weeks, 12 weeks, 6 months, 1 year
Change in strength (N) | Baseline, 6 weeks, 12 weeks, 6 months, 1 year
Change in Simple Shoulder Test9 | Baseline, 6 weeks, 12 weeks, 6 months, 1 year
  The Simple Shoulder Test9 is a self-reported patient outcome score that has been specifically validated to examine post-operative rotator cuff repair outcomes.
Change in American Shoulder and Elbow Surgeon (ASES) Shoulder Score | Baseline, 6 weeks, 12 weeks, 6 months, 1 year
  The ASES Shoulder Score (ref 12) is a self-reported patient outcome score that has been specifically validated to examine rotator cuff disease outcomes. Minimal clinically important differences and the minimal detectable change have been determined.
Change in Marx Shoulder Activity Score2 | Baseline, 6 weeks, 12 weeks, 6 months, 1 year
  The Marx Shoulder Activity Score2 is a validated, patient self-reported outcome score that determines activity level. This is a supplement to outcome scores that measure pain and function.
Change in Single Assessment Numeric Evaluation (SANE) rating | Baseline, 6 weeks, 12 weeks, 6 months, 1 year
  The SANE rating (ref 15) is a simple patient self-reported outcome score that asks the patient to rate their shoulder as a percentage of normal (range 0 to 100%).

CONTACTS AND LOCATIONS:
Overall Officials: Keith M Baumgarten, MD, Principal Investigator — Orthopedic Institute
Locations (1):
- Orthopedic Institute, Sioux Falls, South Dakota, United States

REFERENCES:
- [Derived] Baumgarten KM, Osborn R, Schweinle WE Jr, Zens MJ, Helsper EA. Are Pulley Exercises Initiated 6 Weeks After Rotator Cuff Repair a Safe and Effective Rehabilitative Treatment? A Randomized Controlled Trial. Am J Sports Med. 2016 Jul;44(7):1844-51. doi: 10.1177/0363546516640763. Epub 2016 Apr 26. PMID 27159310